CLINICAL TRIAL: NCT03948997
Title: The Role of Angiogenesis-related Pathways in the Development of Refractory Port Wine Stains
Brief Title: The Role of Angiogenesis-related Pathways in the Development of Port Wine Stains
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: xjpfW (Other)
Collaborators: Air Force General Hospital of the PLA (Other Government); First Hospital of China Medical University (Other); Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor-Investigator, xjpfW, Head of Dermatology, Xijing Hospital
Organization: Xijing Hospital (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: XijingH-PF-20150902
Record Dates: First submitted 2019-05-10; First posted 2019-05-14 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Port Wine Stain
Keywords: port wine stain, PI3K, vascular malformation,PDL
MeSH Terms: conditions — Port-Wine Stain; Hereditary Sensory and Autonomic Neuropathies | interventions — Lasers, Dye

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Patients with port wine stains receive PDL (1.5-10ms, 11-12.5J/cm2) with a treatment range of approximately 10*10cm2
  Interventions: Radiation: Pulsed dye laser (PDL)
- No treatment group (No Intervention): Patients with port wine stains have not been treated with PDL treatment

INTERVENTIONS:
Radiation: Pulsed dye laser (PDL) — Pulsed dye laser (PDL, 595nm) is effective for vasodilatory diseases, especially for the superficial to middle layers of the dermis
  Arms: Treatment group

SUMMARY:
1. Port wine stain (PWS) is a congenital, progressive vascular malformation of human skin involving the superficial vascular plexus that occurs in estimated 3-5 children per 1,000 live births. In childhood, PWS are flat red macules, but lesions tend to darken progressively to purple and, by middle age, often become raised as a result of the development of vascular nodules. Because most malformations occur on the face, PWS is a clinically significant problem in the majority of patients.
2. The late-stage cobblestoning appearance of PWS subjects is comprised by not only pronounced vascular ectasia with proliferation of thin and/or thick-walled vessels and their stroma, but also numerous epithelial, neural and mesenchymal hamartomatous abnormalities. Despite these histologic observations, the specific mechanisms involved in PWS nodular formation remains unclear.
3. In one nodular PWS subject, we found that phosphatidylinositol 3-kinases (PI3K)/protein kinase B (AKT) and phosphoinositide phospholipase C g subunit (PLC-g) were activated in both hypertrophic areas and nodules within the lesion. These observations led us to hypothesize that the PI3K pathway may play an important role in nodular formation.

ELIGIBILITY:
Inclusion Criteria:

* Age 1 month - 70 years old, male or female;
* The patient and the family of the child agreed to participate in the experiment and signed an informed consent form;
* Clinical diagnosis of refractory port wine stains with thickened nodular or PDL resistance; .There is no bleeding, ulceration, infection, etc. affecting the visual field of laser surgery operation.

Exclusion Criteria:

* Patients with severe infectious diseases;
* Heart disease patients;
* Epilepsy patient;
* Pregnant patient;
* Researchers believe that patients who are not suitable for this experiment

Ages: 1 Month to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2015-10-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Exon mutation sequences and mutation frequencies | Baseline (before treatment)
  In patients with nodular port wine stains, the exon mutation sequence and mutation frequency were compared between normal skin tissue (or blood), erythema and nodular tissue of the same patient.

SECONDARY OUTCOMES:
Changes in the levels of cytokines in serum and skin tissues | baseline (before treatment) and 1, 3, 7 days after treatment
  Changes in the levels of VEGF, FGF, HGF, PDGF, TGF-beta and other factors in serum and skin tissues before and after laser treatment

CONTACTS AND LOCATIONS:
Overall Officials: Gang Wang, Prof, Principal Investigator — Dermatology Derpartment of Xijing Hospital

IPD SHARING:
Plan to Share IPD: No